Cover page

Title: Safety and Efficacy of CO2 for Endoscopy

NCT 03287687

12/1/2017

## STATISTICAL ANALYSIS PLAN

Cohort demographics were analyzed using descriptive statistics. Continuous variables were summarized using the mean, and standard deviation (SD) or median and interquartile range (IQR) and compared using the Student t-test for normally-distributed data and the Wilcoxon rank-sum test for data with skewed distribution. Categorical variables were summarized using counts and frequency as a percentage and compared using Chi-Square test or Fisher's exact test. A p-value <0.05 was considered statistically significant. Statistical analysis was performed with SAS 9 statistical software (SAS Institute, Cary, NC).

## Power calculation

The number of subjects enrolled was based on other studies, with the assumption that up to 20% of patients in the air insufflation group would report some degree of abdominal pain after endoscopy. We estimated that the frequency of reported abdominal pain in the CO2 group would be one-fourth of that (5%) seen in the air group. To accomplish this, a minimum total of 150 subjects would be needed (significance level of 5%, power of 80%) so we aimed to recruit a total of 180 patients (enrollment ratio of 1).